CLINICAL TRIAL: NCT06009549
Title: Engagement Trends in Clinical Trials for Metastatic Prostate Cancer - A Journey Into Participation Patterns Among Individuals Affected by the Condition
Brief Title: A Journey Into Participation Patterns Among Metastatic Prostate Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 88079658
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Prostate Cancer
Keywords: metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Taking part in clinical trials usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This research will admit a wide range of data on the clinical study experience of metastatic prostate cancer patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future patients with metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Diagnosis of metastatic prostate cancer
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Enrolled in another research study
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Inability to provide written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with metastatic prostate cancer who are actively considering enrolling in a clinical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to participate in a metastatic prostate cancer clinical research | 3 months
Rate of patients who remain in metastatic prostate cancer clinical research to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pouliot F, Beauregard JM, Saad F, Trudel D, Richard PO, Turcotte E, Rousseau E, Probst S, Kassouf W, Anidjar M, Camirand Lemyre F, Bouvet GF, Neveu B, Tetu A, Guerin B. The Triple-Tracer strategy against Metastatic PrOstate cancer (3TMPO) study protocol. BJU Int. 2022 Sep;130(3):314-322. doi: 10.1111/bju.15621. Epub 2021 Nov 11. PMID 34674367
- [Background] Vlaming M, Bleiker EMA, van Oort IM, Kiemeney LALM, Ausems MGEM. Mainstream germline genetic testing in men with metastatic prostate cancer: design and protocol for a multicenter observational study. BMC Cancer. 2022 Dec 30;22(1):1365. doi: 10.1186/s12885-022-10429-2. PMID 36581909
- [Background] Presti J Jr, Alexeeff S, Horton B, Prausnitz S, Avins AL. Changes in Prostate Cancer Presentation Following the 2012 USPSTF Screening Statement: Observational Study in a Multispecialty Group Practice. J Gen Intern Med. 2020 May;35(5):1368-1374. doi: 10.1007/s11606-019-05561-y. Epub 2019 Dec 9. PMID 31820217

DOCUMENTS (1):
  • Informed Consent Form (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT06009549/ICF_000.pdf